CLINICAL TRIAL: NCT01674686
Title: A Prospective, Single-center, Randomized Study to Evaluate the Effect of Sarpogrelate, a Selective Serotonin Receptor Antagonist, and High Dose Statin on the Reduction of Coronary Spasm in the Patients With Variant Angina
Brief Title: The Effect of Sarpogrelate and High Dose Statin on the Reduction of Coronary Spasm
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, professor, Samsung Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-12-069
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Variant Angina
Keywords: Vasospasm; Sarpogrelate; Statin
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — sarpogrelate; Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Sarpogrelate versus placebo
  Interventions: Drug: Sarpogrelate
- B (Experimental): Atorvastatin 80mg versus no statin or simvastatin 20 mg if LDL > 130 mg/dl
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Sarpogrelate — Sarpogrelate 100mg twice a day
  Arms: A
Drug: Atorvastatin — Atorvastatin 80mg daily
  Arms: B

SUMMARY:
The aim of the study was to to evaluate the effect of sarpogrelate, a selective serotonin receptor antagonist, and high dose statin on the reduction of coronary spasm in the patients with variant angina.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of chest pain compatible with variant angina; morning chest pain aggravated by cold exposure.
* Angiographically proven coronary spasm; TIMI flow < 3 by spontaneous coronary spasm or intracoronary ergonovine spasm provocation test.

Exclusion Criteria:

* Cardiac arrest by coronary spasm
* Left main coronary spasm
* Significant fixed coronary artery stenosis; Diameter stenosis > 70% in the major epicardial artery by coronary angiography
* Left ventricular ejection fraction < 30%
* Coagulation disorders or bleeding tendency (Platelet count < 50k, PT INR > 2.0)
* Significant liver disease (AST or ALT > 100 U/ml)
* Renal failure (S-Cr > 2.0 mg/dl)
* hypersensitivity for statin
* Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Ergonovine provocation test 12months later | 1 year later

SECONDARY OUTCOMES:
C-reactive protein lever 12months later | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hyoen-Cheol Gwon, MD,PhD, Seoul, South Korea